CLINICAL TRIAL: NCT01654250
Title: A Multicenter, Dose-optimized, Double-blind, Randomized, Placebo-controlled Study To Evaluate The Efficacy Of Nwp09 In Pediatric Patients With Attention Deficit Hyperactivity Disorder (Adhd) In A Laboratory Classroom
Brief Title: NWP09 in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NWP09-ADHD-300; B7491005 (Other: Alias Study Number)
Record Dates: First submitted 2012-04-27; First posted 2012-07-31 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; methylphenidate extended-release
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): NWP09
  Interventions: Drug: NWP09
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NWP09 — Methylphenidate, variable dose, daily dosing, 1 week duration
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The safety and efficacy of a chewable formulation of extended-release methylphenidate will be studied in children with ADHD

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years with ADHD who require pharmacologic treatment for this condition

Exclusion Criteria:

* Other serious illnesses or conditions that would put the patient at particular risk for safety events or would interfere with treatment/assessment of ADHD

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Laboratory School, Huntington Beach, California
  - UC Irvine Child Development Center, Irvine, California
  - UC Irvine - Hewitt Hall, Irvine, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Woodland Community Church (Laboratory School), Bradenton, Florida
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Ltd., Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas

REFERENCES:
- [Derived] Wigal SB, Childress A, Berry SA, Belden H, Walters F, Chappell P, Sherman N, Orazem J, Palumbo D. Efficacy and Safety of a Chewable Methylphenidate Extended-Release Tablet in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2017 Oct;27(8):690-699. doi: 10.1089/cap.2016.0177. Epub 2017 May 30. PMID 28557548
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NWP09-ADHD-300&StudyName=NWP09%20in%20Children%20with%20Attention%20Deficit%20Hyperactivity%20Disorder%20%28ADHD%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 90 participants were enrolled in this study, out of which 86 participants were randomized.
Pre-assignment Details: The study consisted of an open-label (OL) dose-optimization phase (1 to 6 weeks), and a placebo-controlled, double blind (DB) for 1 week with no dose adjustments.
Groups:
- Placebo (OL Phase; DB Phase): Placebo-matched to NWP09 chewable tablet once daily optimized dose (optimized during the 1 to 6 weeks OL phase at a starting dose of 20 milligram [mg] and titrated at 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg per day) for 1 week.
- NWP09 (OL Phase; DB Phase): NWP09 chewable tablet once daily optimized dose (optimized during the 1 to 6 weeks OL phase at a starting dose of 20 mg and titrated at 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg per day) for 1 week.
Period: Overall Study
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Started | 44 | 42
Completed | 43 | 42
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who received at least 1 dose of double-blind study medication (either NWP09 or matching placebo) and had at least 1 post-baseline assessment of the primary efficacy variable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase) | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.62) | 9.9 (1.71) | 9.6 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 23 | 30 | 53

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Kotin, Agler, M-Flynn, and Pelham Rating Scale (SKAMP)-Combined Scores-Average of All Post-Dose Time-Points
Description: The SKAMP scale measured the manifestations of attention deficit hyperactivity disorder (ADHD) using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score comprised of 13 items (including subscales: attention with items 1-4, deportment with items 5-8, quality of work with items 9-11 and compliance with items 12-13). The SKAMP composite score was obtained by summing up each item score where each item was rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for a total possible combined score of 0 to 78; where higher score signified worst impairment. Average of all post dose SKAMP-combined scores measured at 0.75, 2, 4, 8, 10, 12 and 13 hours post-dose was calculated.
Time Frame: 0.75 up to 13 hours post-dose
Population: ITT population included all randomized participants who received at least 1 dose of double-blind study medication (either NWP09 or matching placebo) and had at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Number analyzed (Participants) | 43 | 42
units on a scale | 19.1 (1.39) | 12.1 (1.41)
Statistical Analysis 1: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point, and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Square(LS) Mean Difference = -7.0, 95% CI 2-sided [-10.9 to -3.1], Standard Error of Mean 1.99

2. Secondary Outcome: Onset and Duration of Clinical Effect
Description: Onset and duration of clinical effect was determined using SKAMP combined rating scale at each post-dose time point. Onset of effect was defined as first assessment time showing statistical significance (i.e. p was less than or equal to [=<] 0.05) between NWP09 and placebo and duration of effect was defined as the as last consecutive time-point at which difference was statistically significant between NWP09 and placebo. SKAMP scale measured the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. SKAMP combined score was comprised of 13 items [subscales: attention (1-4 items), deportment (5-8 items), quality of work (9-11 items) and compliance (12-13 items)]. SKAMP combined score was obtained by summing up each item score where each item was rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 78; where higher score signified worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12, 13 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Number analyzed (Participants) | 43 | 42
Units on a scale
  Hour 0.75 | 18.3 (11.21) | 10.7 (9.79)
  Hour 2 | 20.3 (13.11) | 8.0 (6.88)
  Hour 4 | 19.8 (12.99) | 8.1 (6.74)
  Hour 8 | 19.3 (11.34) | 12.1 (10.38)
  Hour 10 | 17.7 (11.58) | 14.8 (10.26)
  Hour 12 | 19.4 (11.23) | 17.0 (12.79)
  Hour 13 | 18.4 (10.73) | 17.5 (13.38)
Statistical Analysis 1: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -8.2, 95% CI 2-sided [-12.7 to -3.7], Standard Error of Mean 2.28
Statistical Analysis 2: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose: Adjusted p-values were generated using a fixed sequence testing procedure from p-values which were generated from the mixed effects model; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.8, 95% CI 2-sided [-17.3 to -8.3], Standard Error of Mean 2.28
Statistical Analysis 4: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose: Adjusted p-values were generated using a fixed sequence testing procedure from p-values which were generated from the mixed effects model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.3, 95% CI 2-sided [-16.8 to -7.8], Standard Error of Mean 2.28
Statistical Analysis 6: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose: Adjusted p-values were generated using a fixed sequence testing procedure from p-values which were generated from the mixed effects model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effect and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.8, 95% CI 2-sided [-12.3 to -3.3], Standard Error of Mean 2.28
Statistical Analysis 8: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose: Adjusted p-values were generated using a fixed sequence testing procedure from p-values which were generated from the mixed effects model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 post-dose: Nominal p-value -treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; LS Mean Difference = -3.4, 95% CI 2-sided [-7.9 to 1.1], Standard Error of Mean 2.28
Statistical Analysis 10: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 post-dose: Adjusted p-value were generated using a fixed sequence testing procedure from p-values generated from the mixed effects model; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.206, Mixed Models Analysis; LS Mean Difference = -2.9, 95% CI 2-sided [-7.4 to 1.6], Standard Error of Mean 2.28
Statistical Analysis 12: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose: Adjusted p-values are generated using a fixed sequence testing procedure from p-values which were generated from the mixed effects model; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis
Statistical Analysis 13: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose: Nominal p value-treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.496, Mixed Models Analysis; LS Mean Difference = -1.6, 95% CI 2-sided [-6.0 to 2.9], Standard Error of Mean 2.28
Statistical Analysis 14: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose: Adjusted p-value were generated using a fixed sequence testing procedure from p-values generated from the mixed effects model; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis

3. Secondary Outcome: Swanson, Kotin, Agler, M-Flynn, and Pelham Rating Scale (SKAMP) SKAMP Attention and Deportment Subscale Scores at Hour 0.75, 2, 4, 8, 10, 12 and 13 Post-Dose
Description: SKAMP scale measured the manifestations of ADHD using an independent observer rating of the participant's impairment in classroom observed behaviors. The SKAMP subscales were obtained by summing the individual items as follows: Attention (items 1-4) and Deportment (items 5-8), where each item was rated on a 7-point scale (0=normal to 6=maximal impairment). SKAMP attention subscale was reported which evaluates concentration in the classroom and comprises of 4 items, with a total possible score for of 0 to 24; higher score indicates worst impairment. SKAMP deportment subscale was reported which assesses behavior in the classroom and comprises of 4 items, with a total possible score for each sub-scale of 0 to 24; higher score indicates worst impairment.
Time Frame: 0.75, 2, 4, 8, 10, 12, 13 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Number analyzed (Participants) | 43 | 42
Units on a scale
  Hour 0.75: Attention Subscale | 2.9 (2.72) | 1.6 (2.35)
  Hour 0.75: Deportment Subscale | 4.6 (4.91) | 2.1 (3.74)
  Hour 2: Attention Subscale | 3.4 (3.27) | 1.1 (1.85)
  Hour 2: Deportment Subscale | 5.4 (5.31) | 1.6 (2.43)
  Hour 4: Attention Subscale | 3.2 (2.92) | 1.0 (1.48)
  Hour 4: Deportment Subscale | 5.4 (5.22) | 1.7 (3.29)
  Hour 8: Attention Subscale | 3.5 (2.92) | 2.0 (2.82)
  Hour 8: Deportment Subscale | 4.3 (4.73) | 2.6 (4.33)
  Hour 10: Attention Subscale | 3.4 (2.70) | 2.6 (3.49)
  Hour 10: Deportment Subscale | 3.9 (4.86) | 2.6 (3.18)
  Hour 12: Attention Subscale | 3.4 (2.91) | 3.2 (3.26)
  Hour 12: Deportment Subscale | 4.2 (4.46) | 3.5 (5.48)
  Hour 13: Attention Subscale | 3.8 (3.15) | 3.2 (3.35)
  Hour 13: Deportment Subscale | 3.7 (4.30) | 3.9 (5.48)
Statistical Analysis 1: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; LS Mean Difference = -1.5, 95% CI 2-sided [-2.6 to -0.4], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.5, 95% CI 2-sided [-3.6 to -1.4], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.3, 95% CI 2-sided [-3.4 to -1.2], Standard Error of Mean 0.56
Statistical Analysis 4: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference = -1.7, 95% CI 2-sided [-2.8 to -0.6], Standard Error of Mean 0.56
Statistical Analysis 5: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.097, Mixed Models Analysis; LS Mean Difference = -0.9, 95% CI 2-sided [-2.0 to 0.2], Standard Error of Mean 0.56
Statistical Analysis 6: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.490, Mixed Models Analysis; LS Mean Difference = -0.4, 95% CI 2-sided [-1.5 to 0.7], Standard Error of Mean 0.56
Statistical Analysis 7: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose attention subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.164, Mixed Models Analysis; LS Mean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.56
Statistical Analysis 8: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose deportment subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = -2.7, 95% CI 2-sided [-4.6 to -0.9], Standard Error of Mean 0.94
Statistical Analysis 9: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose deportment subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean difference = -3.9, 95% CI 2-sided [-5.8 to -2.1], Standard Error of Mean 0.94
Statistical Analysis 10: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose deportment sub scale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -3.9, 95% CI 2-sided [-5.8 to -2.1], Standard Error of Mean 0.94
Statistical Analysis 11: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose deportment subscale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis; LS Mean Difference = -1.9, 95% CI 2-sided [-3.8 to -0.1], Standard Error of Mean 0.94
Statistical Analysis 12: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 post-dose deportment sub scale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.118, Mixed Models Analysis; LS Mean Difference = -1.5, 95% CI 2-sided [-3.3 to 0.4], Standard Error of Mean 0.94
Statistical Analysis 13: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose deportment sub scale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.342, Mixed Models Analysis; LS Mean Difference = -0.9, 95% CI 2-sided [-2.7 to 1.9], Standard Error of Mean 0.94
Statistical Analysis 14: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose deportment sub scale: Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.962, Mixed Models Analysis; LS Mean Difference = 0.0, 95% CI 2-sided [-1.8 to 1.9], Standard Error of Mean 0.94

4. Secondary Outcome: Permanent Product Measure of Performance (PERMP) Scores at Hour 0.75, 2, 4, 8, 10, 12 and 13 Post-Dose
Description: The PERMP score measured the manifestations of attention deficit hyperactivity disorder. The PERMP is a 10-minute written test, on 80 math problems, performed as seatwork in the classroom. At the end of the 10- minute math test , the PERMP score of the number of math problems attempted plus the number of math problems answered correctly in a 10-minute session was used to measure participant's performance. The total score range from 0-160 with higher scores indicating better performance.
Time Frame: 0.75, 2, 4, 8, 10, 12 and 13 post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Number analyzed (Participants) | 43 | 42
Units on a scale
  Hour 0.75: Problems attempted | 105.4 (51.08) | 128.8 (53.32)
  Hour 0.75: Problems corrected | 102.8 (51.62) | 123.9 (55.11)
  Hour 2: Problems attempted | 106.6 (55.22) | 140.9 (57.85)
  Hour 2: Problems corrected | 103.7 (55.75) | 136.6 (60.34)
  Hour 4: Problems attempted | 107.2 (55.89) | 140.0 (62.88)
  Hour 4: Problems corrected | 104.2 (56.72) | 135.6 (64.53)
  Hour 8: Problems attempted | 101.7 (53.32) | 129.1 (62.64)
  Hour 8: Problems corrected | 98.5 (53.71) | 124.0 (63.92)
  Hour 10: Problems attempted | 103.2 (53.54) | 113.9 (62.33)
  Hour 10: Problems corrected | 100.8 (53.99) | 107.9 (63.08)
  Hour 12: Problems attempted | 97.9 (48.86) | 111.1 (55.70)
  Hour 12: Problems corrected | 95.1 (49.25) | 103.3 (57.76)
  Hour 13: Problems attempted | 98.6 (46.01) | 115.4 (57.30)
  Hour 13: Problems corrected | 95.0 (45.76) | 101.8 (58.94)
Statistical Analysis 1: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; LS Mean difference = 25.3, 95% CI 2-sided [3.4 to 47.1], Standard Error of Mean 11.12
Statistical Analysis 2: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = 36.1, 95% CI 2-sided [14.2 to 57.9], Standard Error of Mean 11.12
Statistical Analysis 3: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS Mean Difference = 34.7, 95% CI 2-sided [12.8 to 56.6], Standard Error of Mean 11.12
Statistical Analysis 4: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; LS Mean Difference = 29.3, 95% CI 2-sided [7.4 to 51.1], Standard Error of Mean 11.12
Statistical Analysis 5: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.261, Mixed Models Analysis; LS Mean Difference = 12.5, 95% CI 2-sided [-9.3 to 34.4], Standard Error of Mean 11.12
Statistical Analysis 6: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; LS Mean Difference = 15.1, 95% CI 2-sided [-6.7 to 37.0], Standard Error of Mean 11.12
Statistical Analysis 7: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose (Problems attempted): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.094, Mixed Models Analysis; LS Mean Difference = 18.7, 95% CI 2-sided [-3.2 to 40.5], Standard Error of Mean 11.12
Statistical Analysis 8: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 0.75 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis; LS Mean Difference = 22.6, 95% CI 2-sided [0.1 to 45.1], Standard Error of Mean 11.44
Statistical Analysis 9: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 2 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference = 34.4, 95% CI 2-sided [11.9 to 56.9], Standard Error of Mean 11.44
Statistical Analysis 10: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 4 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = 32.9, 95% CI 2-sided [10.5 to 55.4], Standard Error of Mean 11.44
Statistical Analysis 11: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 8 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; LS Mean Difference = 27.0, 95% CI 2-sided [4.5 to 49.5], Standard Error of Mean 11.44
Statistical Analysis 12: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 10 (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.451, Mixed Models Analysis; LS Mean difference = 8.6, 95% CI 2-sided [-13.9 to 31.1], Standard Error of Mean 11.44
Statistical Analysis 13: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 12 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.394, Mixed Models Analysis; LS Mean Difference = 9.8, 95% CI 2-sided [-12.7 to 32.2], Standard Error of Mean 11.44
Statistical Analysis 14: Comparison: Placebo (OL Phase; DB Phase) vs NWP09 (OL Phase; DB Phase); Hour 13 post-dose (Problems correct): Treatment comparisons for observed scores were assessed using a mixed model repeated measures analysis, with treatment (NWP09/Placebo), study center, time point and time point by treatment interaction as main effects and participant intercept as a random effect; Test type: Superiority or Other; p = 0.466, Mixed Models Analysis; LS Mean difference = 8.3, 95% CI 2-sided [-14.1 to 30.8], Standard Error of Mean 11.44

5. Other Pre Specified Outcome: Clinical Global Impression of Severity (CGI-S)
Description: CGI-S scale was used to measure features associated with ADHD. The assessment was performed by the investigator of the study research team. The CGI-S classified the participant's current disease status as: 1 = normal, not at all ill, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = among the most extremely ill participants. This outcome measure was analyzed during open label phase in entire study population prior to randomization into two treatment groups.
Time Frame: Baseline, Day 8, 15, 22, 29, 36, 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Entire Study Population: All randomized participants received either placebo-matched to NW09 or NW09 chewable tablets once daily optimized dose (optimized during the 4 to 6 weeks open label phase at a starting dose of 20 mg and titrated at 10 or 20 mg increments, based on clinical response and tolerability to a maximum daily dose of 60 mg per day) for 1 week.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 85
Units on a scale
  Baseline | 4.6 (0.66)
  Day 8 | 3.9 (1.29)
  Day 15 | 3.3 (1.16)
  Day 22 | 2.6 (1.05)
  Day 29 | 2.2 (1.02)
  Day 36 | 2.0 (0.82)
  Day 43 | 2.0 (0.89)

6. Other Pre Specified Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: The CGI-I measured the participant's disease improvement relative to baseline as followed: 1= very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6= much worse, and 7=very much worse. This outcome measure was analyzed during open label phase in entire study population prior to randomization into two treatment groups.
Time Frame: Day 8, 15, 22, 29, 36, 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Entire Study Population
Number analyzed (Participants) | 85
Units on a scale
  Day 8 | 3.0 (1.07)
  Day 15 | 2.3 (0.94)
  Day 22 | 1.7 (0.69)
  Day 29 | 1.4 (0.56)
  Day 36 | 1.3 (0.49)
  Day 43 | 1.3 (0.46)

7. Other Pre Specified Outcome: Conners Parent Rating Scale (CPRS) Scores
Description: CPRS was used to measure features associated with ADHD and was used to compare scores during the dose optimization period i.e. 1-6 weeks. The assessment was performed by parent or guardian. CPRS consisted of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true). Raw scores were converted to t-scores and t-scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. The participant received normalized t-scores on the following scales: oppositional, cognitive problems/inattention, hyperactivity, anxious-shy, perfectionism, social problems, psychosomatic, ADHD index, restless-impulse, emotional liability, conner's global index, inattentive, hyperactive-impulsive and diagnostic and statistical manual of mental disorders IV (DSM-IV). This outcome measure was analyzed during open label phase in entire study population prior to randomization into two treatment groups.
Time Frame: Baseline, Day 8, 15, 22, 29, 36, 43
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Entire Study Population
Number analyzed (Participants) | 85
Units on a scale
  Oppositional : Baseline | 67.3 (15.08)
  Cognitive Problems/ Inattention: Baseline | 71.1 (13.30)
  Hyperactivity: Baseline | 79.3 (16.18)
  Anxious-shy: Baseline | 57.3 (15.06)
  Perfectionism: Baseline | 54.9 (12.75)
  Social problems: Baseline | 57.1 (14.31)
  Psychosomatic: Baseline | 57.1 (17.63)
  ADHD index: Baseline | 73.8 (11.00)
  Restless-Impulse: Baseline | 74.6 (12.48)
  Emotional Liability: Baseline | 64.8 (15.82)
  Conner's Global index: Baseline | 73.6 (13.25)
  Inattentive: Baseline | 73.8 (12.57)
  Hyperactive-Impulsive: Baseline | 78.0 (14.43)
  DSM-IV: Baseline | 77.8 (12.04)
  Oppositional: Day 8 | 64.0 (15.89)
  Cognitive Problems/ Inattention: Day 8 | 66.5 (13.33)
  Hyperactivity: Day 8 | 73.5 (17.81)
  Anxious-shy: Day 8 | 54.9 (13.99)
  Perfectionism: Day 8 | 52.7 (11.80)
  Social problems: Day 8 | 55.5 (13.06)
  Psychosomatic: Day 8 | 55.2 (17.22)
  ADHD index: Day 8 | 68.8 (13.30)
  Restless-Impulse: Day 8 | 69.7 (14.51)
  Emotional Liability: Day 8 | 62.1 (15.25)
  Conner's Global index: Day 8 | 68.9 (15.06)
  Inattentive: Day 8 | 68.3 (13.46)
  Hyperactive-Impulsive: Day 8 | 73.1 (16.24)
  DSM-IV: Day 8 | 72.1 (14.62)
  Oppositional: Day 15 | 59.5 (14.75)
  Cognitive Problems/ Inattention: Day 15 | 61.8 (12.88)
  Hyperactivity: Day 15 | 68.0 (17.58)
  Anxious-shy: Day 15 | 52.5 (13.55)
  Perfectionism: Day 15 | 51.1 (11.51)
  Social problems: Day 15 | 54.0 (12.71)
  Psychosomatic: Day 15 | 53.2 (15.93)
  ADHD index: Day 15 | 63.3 (12.70)
  Restless-Impulse: Day 15 | 65.2 (13.96)
  Emotional Liability: Day 15 | 57.0 (13.84)
  Conner's Global index: Day 15 | 63.6 (14.08)
  Inattentive: Day 15 | 63.0 (13.39)
  Hyperactive-Impulsive: Day 15 | 67.4 (15.86)
  DSM-IV: Day 15 | 66.2 (14.33)
  Oppositional: Day 22 | 55.5 (13.27)
  Cognitive Problems/ Inattention: Day 22 | 59.1 (12.30)
  Hyperactivity: Day 22 | 62.8 (14.73)
  Anxious-shy: Day 22 | 50.5 (12.66)
  Perfectionism: Day 22 | 49.3 (10.08)
  Social problems: Day 22 | 52.6 (12.65)
  Psychosomatic: Day 22 | 50.6 (14.54)
  ADHD index: Day 22 | 59.7 (12.18)
  Restless-Impulse: Day 22 | 59.6 (12.86)
  Emotional Liability: Day 22 | 53.3 (12.60)
  Conner's Global index: Day 22 | 58.4 (13.17)
  Inattentive: Day 22 | 59.5 (12.44)
  Hyperactive-Impulsive: Day 22 | 63.5 (14.48)
  DSM-IV: Day 22 | 62.3 (13.30)
  Oppositional: Day 29 | 52.8 (11.28)
  Cognitive Problems/ Inattention: Day 29 | 55.7 (10.97)
  Hyperactivity: Day 29 | 58.2 (12.87)
  Anxious-shy: Day 29 | 49.8 (12.08)
  Perfectionism: Day 29 | 48.3 (9.63)
  Social problems: Day 29 | 51.2 (10.40)
  Psychosomatic: Day 29 | 49.7 (12.13)
  ADHD index: Day 29 | 55.7 (9.88)
  Restless-Impulse: Day 29 | 55.9 (10.77)
  Emotional Liability: Day 29 | 51.0 (10.29)
  Conner's Global index: Day 29 | 54.8 (10.88)
  Inattentive: Day 29 | 55.6 (11.19)
  Hyperactive-Impulsive: Day 29 | 57.8 (12.08)
  DSM-IV: Day 29 | 57.1 (11.10)
  Oppositional: Day 36 | 50.5 (10.42)
  Cognitive Problems/ Inattention: Day 36 | 54.7 (11.44)
  Hyperactivity: Day 36 | 56.0 (12.36)
  Anxious-shy: Day 36 | 49.0 (10.90)
  Perfectionism: Day 36 | 46.6 (8.08)
  Social problems: Day 36 | 50.1 (10.10)
  Psychosomatic: Day 36 | 47.9 (10.37)
  ADHD index: Day 36 | 53.8 (10.15)
  Restless-Impulse: Day 36 | 54.3 (10.79)
  Emotional Liability: Day 36 | 49.8 (9.76)
  Conner's Global index: Day 36 | 53.3 (10.90)
  Inattentive: Day 36 | 54.7 (11.49)
  Hyperactive-Impulsive: Day 36 | 55.2 (11.15)
  DSM-IV: Day 36 | 55.4 (10.96)
  Oppositional: Day 43 | 49.8 (10.81)
  Cognitive Problems/ Inattention: Day 43 | 54.0 (11.48)
  Hyperactivity: Day 43 | 54.4 (10.63)
  Anxious-shy: Day 43 | 47.9 (10.80)
  Perfectionism: Day 43 | 45.9 (7.60)
  Social problems: Day 43 | 50.5 (10.77)
  Psychosomatic: Day 43 | 47.2 (9.87)
  ADHD index: Day 43 | 52.9 (9.84)
  Restless-Impulse: Day 43 | 53.2 (10.37)
  Emotional Liability: Day 43 | 48.9 (9.21)
  Conner's Global index: Day 43 | 52.1 (10.16)
  Inattentive: Day 43 | 53.8 (11.14)
  Hyperactive-Impulsive: Day 43 | 54.3 (10.30)
  DSM-IV: Day 43 | 54.3 (10.74)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo (OL Phase; DB Phase) | NWP09 (OL Phase; DB Phase)
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 31/44 | 33/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (OL Phase; DB Phase) (N=44) | NWP09 (OL Phase; DB Phase) (N=42)
Decreased appetite (Metabolism and nutrition disorders) | 17 | 15
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 4 | 8
Insomnia (Psychiatric disorders) | 7 | 2
Initial insomnia (Psychiatric disorders) | 3 | 2
Middle insomnia (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 0 | 1
Anger (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Change in sustained attention (Psychiatric disorders) | 1 | 0
Emotional poverty (Psychiatric disorders) | 0 | 1
Onychophagia (Psychiatric disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 7
Viral infection (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Streptococcal impetigo (Infections and infestations) | 1 | 0
Tic (Psychiatric disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 3
Dysgeusia (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 1 | 1
Aphonia (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Irritability (General disorders) | 6 | 5
Feeling jittery (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
Malaise (General disorders) | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Excessive eye blinking (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Blood pressure systolic increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Enuresis (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.